CLINICAL TRIAL: NCT00462982
Title: A Phase II Study of SU11248 (Sunitinib) in Patients With Renal Cell Carcinoma and Melanoma Metastatic to the Brain
Brief Title: Sunitinib in Treating Patients With Brain Metastases Caused by Kidney Cancer or Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-009; P30CA008748 (NIH); MSKCC-07009
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-11

CONDITIONS: Kidney Cancer; Melanoma (Skin); Metastatic Cancer
Keywords: stage IV melanoma; tumors metastatic to brain; stage IV renal cell cancer; recurrent melanoma; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Neoplasm Metastasis; Brain Neoplasms; Carcinoma, Renal Cell | interventions — Sunitinib

ARMS (1):
- Sunitinib (Experimental): Patients will be treated with 50 mg daily for four out of every six weeks.
  Interventions: Drug: sunitinib malate

INTERVENTIONS:
Drug: sunitinib malate

SUMMARY:
RATIONALE: Sunitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well sunitinib works in treating patients with brain metastases caused by kidney cancer or melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of sunitinib malate, in terms of objective radiographic response of brain lesions, in patients with brain metastases secondary to renal cell carcinoma or melanoma.

Secondary

* Determine overall and progression-free survival.

OUTLINE: Patients receive oral sunitinib malate once daily on days 1-28. Courses repeat every 6 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed melanoma or renal cell carcinoma

  * Metastatic brain disease
* Must have assessable target intracranial lesion(s), defined as measurable disease ≥ 10 mm in longest diameter that is not appropriate for stereotactic radiosurgery or surgical resection

  * Lesions previously treated with radiosurgery AND not eligible for resection can only be used as target lesions if there has been true tumor progression on baseline scan (i.e., ≥ 20% increase in longest diameter of lesion) rather than radionecrosis

    * True progression must be confirmed by PET scan or other corroborating imaging used to distinguish radionecrosis
* No leptomeningeal metastases or primary dural metastases

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky PS 60-100%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Total leukocyte count ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 2.0 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Hemoglobin ≥ 9.0 g/dL
* Calcium ≤ 12.0 mg/dL
* AST and ALT ≤ 1.5 times ULN
* PT ≤ 1.5 times ULN
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No uncontrolled medical illness including, but not limited to, any of the following:

  * Hypertension (i.e., blood pressure > 150/100 mm Hg)
  * Thyroid disease
  * Severe valvular disease
  * Severe pulmonary disease
  * HIV/AIDS
  * Severe psychiatric illness
* No cardiac dysrhythmia ≥ grade 2
* No prolonged QTc interval on baseline EKG
* No systemic hemorrhage ≥ grade 2 within the past 4 weeks

  * No CNS hemorrhage ≥ grade 2

    * Grade 1 (asymptomatic) CNS hemorrhage allowed at investigator's discretion
* None of the following within the past 6 months:

  * Myocardial infarction
  * Unstable angina
  * Symptomatic congestive heart failure
  * Stroke/transient ischemic attack
  * Pulmonary embolism
* Ejection fraction ≥ 50% by baseline echocardiogram OR < 20% decrease in ejection fraction from a prior study

PRIOR CONCURRENT THERAPY:

* No prior multi-targeted tyrosine kinase inhibitor therapy (e.g., sunitinib malate or sorafenib)
* No coronary/peripheral arterial bypass surgery within the past 6 months
* More than 4 weeks since prior surgery and recovered
* More than 4 weeks since prior and no other concurrent experimental therapy or cytotoxic chemotherapy
* More than 4 weeks since prior immunotherapy
* More than 2 weeks since prior stereotactic radiosurgery and recovered
* More than 7 days since prior and no concurrent drugs that interact with CYP3A4 family, including enzyme-inducing antiepileptic drugs, warfarin, or Hypericum perforatum extract (St. John's wort)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-03; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren E. Abrey, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Paul B. Chapman, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Robert J. Motzer, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sunitinib
Started | 8
Completed | 5
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Patient Not Treated | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Central Nervous System (CNS) Response Rate by RECIST Criteria
Description: Response and progression will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in RECIST. Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques (CT, MRI, X-ray) or as >10 mm with spiral CT scan. This study will use a minimum diameter of 10 mm for measurable lesions in the brain, regardless of imaging modality. All tumor measurements must be recorded in millimeters (or decimal fractions of centimeters). All other lesions are considered non-measurable disease. Bone lesions, leptomeningeal disease, ascites, pleural/pericardial effusions, inflammatory breast disease, and cystic lesions are all nonmeasurable.
Time Frame: up to a year
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 5
participants
  Stable Disease (SD) | 3
  Progression of Disease (POD) | 2

ADVERSE EVENTS:
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=8)
ALT, SGPT (Blood and lymphatic system disorders) | 1 (1)
AST, SGOT (Blood and lymphatic system disorders) | 1 (1)
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 1 (1)
Pain - Head/headache (General disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Speech impairment (Nervous system disorders) | 1 (1)
Thrombosis/thrombus/embolism (Cardiac disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib (N=8)
ALT, SGPT (Blood and lymphatic system disorders) | 1 (1)
AST, SGOT (Blood and lymphatic system disorders) | 1 (1)
Albumin, low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 3 (3)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (1)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes